CLINICAL TRIAL: NCT01517802
Title: A Phase 3b Multicenter, Open-label Abiraterone Acetate Long-term Safety Study
Brief Title: A Study That Provides Long-term Safety Follow-up and Examines Long-term Exposure to Abiraterone Acetate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100797; 212082PCR3010 (Other: Janssen Research & Development, LLC); 2011-005243-28 (EudraCT Number)
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Metastatic Breast Cancer
Keywords: Metastatic castration-resistant prostate cancer; Metastatic breast cancer; Abiraterone acetate; Low-dose corticosteroid treatment; Long-term access
MeSH Terms: conditions — Breast Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): Patients will continue the same treatment regimen they were receiving during their participation in the previous abiraterone acetate clinical study.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Type=exact number, unit=mg, number=1000, form=tablet, route=oral, abiraterone acetate once daily
Drug: Prednisone — Type=exact number, unit=mg, number=5, form=tablet, route=oral, prednisone or prednisolone twice daily

SUMMARY:
The purpose of this study is to collect follow-up safety data from participants in completed abiraterone acetate studies for a maximum duration of 9 years.

DETAILED DESCRIPTION:
This is a nonrandomized (individuals will not be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), long-term safety follow-up study of abiraterone acetate in approximately 300 patients from other completed abiraterone acetate clinical studies. Patients must have received at least 3 months of treatment with abiraterone acetate and a low-dose corticosteroid and, based on investigator assessment, may benefit from continued treatment. This study will consist of a screening period followed by open-label treatment of continued abiraterone acetate access. The patients will continue with the same abiraterone acetate and low-dose corticosteroid dosing regimen they were receiving in the previous abiraterone acetate clinical study until the investigator determines that the patient is no longer receiving benefit or the sponsor terminates the study. Patients can be withdrawn from the study if an alternative access (eg, patient-assistance program or commercial source of abiraterone acetate) is available and feasible. Each cycle of treatment will be 28 days. Investigators will monitor and assess the patients for response to treatment or progression according to routine practice or as clinically indicated to determine whether continued treatment with abiraterone acetate is warranted. No efficacy data are being collected. Safety will be monitored throughout the study for a maximum duration of 9 years. End-of-study assessments will be performed at least 30 days after the last dose of abiraterone or upon early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in an abiraterone acetate clinical study considered complete and had received at least 3 months of treatment with abiraterone acetate tablets.

Exclusion Criteria:

* Medical conditions that require hospitalization.
* Any condition or situation which, in the opinion of the investigator, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (22):
- United States (10):
  - Aurora, Colorado
  - Marrero, Louisiana
  - Boston, Massachusetts
  - Omaha, Nebraska
  - East Setauket, New York
  - New York, New York
  - Myrtle Beach, South Carolina
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Houston, Texas
- Australia (4):
  - Kogarah
  - Kurralta Park
  - South Brisbane
  - Subiaco
- Antwerp, Belgium
- Hamburg, Germany
- Barcelona, Spain
- Uppsala, Sweden
- United Kingdom (4):
  - Newcastle upon Tyne
  - Northwood
  - Sutton
  - Whitchurch

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 32 randomized participants, 1 participant did not receive any dose of drug and hence was excluded from all the analyses.
Groups:
- Abiraterone Acetate + Prednisone/Prednisolone: Participants who received at least 3 months of abiraterone acetate treatment in previously completed abiraterone acetate studies (COU-AA-001 [NCT00473512], COU-AA-002 [NCT00473746], COU-AA-006 [NCT00910754], COU-AA-206 [NCT01400555], COU-AA-301 [NCT00638690], COU-AA-302 [NCT00887198], COU-AA-BMA [NCT00544440]) continued to receive abiraterone acetate 1000 milligrams (mg) (four 250 mg tablets) along with low dose corticosteroid (prednisone/prednisolone) 5 mg tablet orally twice daily starting Day 1 Cycle 1 (each cycle was of 28 days) according to dosing regimen established in the previously completed study until the investigator determined that the participant no longer received benefit or the sponsor terminated the study or the participant had continued the treatment in this study and were followed-up for safety for up to 9 years.
Period: Overall Study
Arm/Group | Abiraterone Acetate + Prednisone/Prednisolone
Started | 31
Completed | 30
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate + Prednisone/Prednisolone
Number analyzed (Participants) | 31
Age, Customized [Count of Participants; unit: Participants]
  63-90 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or is an important medical event.
Time Frame: Up to 9 years
Population: Safety analysis set included participants that received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate + Prednisone/Prednisolone
Number analyzed (Participants) | 31
Participants | 16

ADVERSE EVENTS:
Time Frame: Up to 9 years
Description: Safety analysis set included participants who received at least 1 dose of study drug.
Arm/Group | Abiraterone Acetate + Prednisone/Prednisolone
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 16/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone/Prednisolone (N=31)
Lower Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Aortic Thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Fatigue (General disorders) | 1
Weight Decreased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Skin Laceration (Injury, poisoning and procedural complications) | 2
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Aortic Valve Replacement (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone/Prednisolone (N=31)
Lower Respiratory Tract Infection (Infections and infestations) | 0
Urinary Tract Infection (Infections and infestations) | 0
Dehydration (Metabolism and nutrition disorders) | 0
Cerebrovascular Accident (Nervous system disorders) | 0
Encephalopathy (Nervous system disorders) | 0
Spinal Cord Compression (Nervous system disorders) | 0
Syncope (Nervous system disorders) | 0
Cardiac Failure (Cardiac disorders) | 0
Cardiac Failure Congestive (Cardiac disorders) | 0
Myocardial Infarction (Cardiac disorders) | 0
Aortic Thrombosis (Vascular disorders) | 0
Hypertension (Vascular disorders) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0
Diarrhoea (Gastrointestinal disorders) | 0
Nausea (Gastrointestinal disorders) | 0
Oesophagitis (Gastrointestinal disorders) | 0
Vomiting (Gastrointestinal disorders) | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0
Acute Kidney Injury (Renal and urinary disorders) | 0
Urinary Retention (Renal and urinary disorders) | 0
Fatigue (General disorders) | 0
Weight Decreased (Investigations) | 0
Fall (Injury, poisoning and procedural complications) | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0
Aortic Valve Replacement (Surgical and medical procedures) | 0

LIMITATIONS AND CAVEATS:
No site qualification or initiation visits conducted for previous studies on abiraterone acetate. No formal case report forms were developed nor clinical database was generated to capture data in this study. Due to disease condition, most of participants were lost to follow-up and hence data collected was not as planned. Data were recorded based on available source notes at participating sites and thereby into CIOMS. Studied population was very small hence it was difficult to generalize results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT01517802/Prot_SAP_000.pdf